CLINICAL TRIAL: NCT05531097
Title: A Randomized, Double-blind, Placebo-controlled Study of the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of Single Doses and Multiple Dose of HSK31679 in Healthy Volunteers and Subjects With Elevated LDL-C
Brief Title: Ascending Single-Dose and Multiple-Dose Study to Evaluate HSK31679 in Healthy Subjects and Subjects With Elevated LDL-C
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Haisco Pharmaceutical Group Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: HSK31679-101
Record Dates: First submitted 2022-08-24; First posted 2022-09-07 (Actual); Last update posted 2024-01-03 (Actual); Status verified 2024-01

CONDITIONS: Healthy; Elevated LDL-C
Keywords: HSK31679; Healthy; Elevated LDL-C; Phase I

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HSK31679 (Experimental)
  Interventions: Drug: HSK31679
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: HSK31679 — Single or multiple oral doses of HSK31679
  Arms: HSK31679
Drug: Placebo — Matching placebo
  Arms: Placebo

SUMMARY:
This is a Phase I, single-dose and multiple dose escalation clinical trial for HSK31679 conducted in chinese healthy volunteers and LDL-C elevated subjects. The safety, tolerability, food-impact,pharmacokinetics and pharmacodynamics of HSK31679 tablet in healthy volunteers and LDL-C elevated volunteers will be evaluated using a randomized, double-blind, placebo-controlled trial design

ELIGIBILITY:
Inclusion Criteria:

1. The subject must be willing and able to provide written informed consent.
2. At the time of screening, eligibility criteria for SAD part are 18 to 55 years of age , and eligibility criteria for MAD part are 18 to 60 years of age , both male and female.
3. Body mass index ≥ 18.0 and ≤ 30.0 kg/m2, with a body weight ≥ 45 kg at Screening.
4. LDL cholesterol ≥ 70mg/dL for SAD part and LDL cholesterol ≥ 100mg/dL for MAD part.
5. Triglyceride <400 mg/dL.
6. Medically healthy without clinically significant abnormalities at Screening and predose on Day 1, including:

   1. Physical examination without any clinically relevant findings.
   2. Heart rate in the range of 50 to 100 bpm after 5 minutes rest in supine position or seated.
   3. Body temperature, between 35.0°C and 37.7°C.
   4. Three conventional 12-ECG recordings (the average of the three measurements will be used to determine eligibility) were consistent with normal cardiac conduction and function.
7. Fertile male and female subjects agree to use appropriate physical contraception during the study and for 6 months after the last dose.
8. Willing and able to comply with all study evaluations and adhere to protocol schedules and constraints.
9. Additional inclusion criteria for SAD and MAD subjects who are not treated with statins: Systolic blood pressure in the range of 90 to 139 mmHg and diastolic blood pressure in the range of 60 to 89 mmHg after 5 minutes in supine position or seated.
10. Additional inclusion criteria for MAD subjects who are treated with statins:

    1. Systolic blood pressure in the range of 90 to 160 mmHg and diastolic blood pressure in the range of 60 to 100 mmHg after 5 minutes in supine position or seated.
    2. A stable dose of a statin (simvastatin atorvastatin or rosuvastatin) is administered daily for 28 days before randomization.

Exclusion Criteria:

1. history or presence of major diseases of the cardiovascular, respiratory, digestive, urological, hematologic, endocrine, immunologic, skin or nervous system, as well as any acute illness or surgical procedure within the past 3 months as determined by the investigator to be clinically relevant. Any clinically significant uncontrolled endocrine or immune disease known to affect lipid or lipoprotein levels.
2. Current infection requiring treatment with antibiotics, antifungal, antiparasitic, or antiviral agents.
3. Any history of malignancy within the last 10 years.
4. Previous thyroid related disease and/or abnormal thyroid function tests during screening are clinically significant.
5. Laboratory tests during the screening period were abnormal and clinically significant as judged by the investigator . [The abnormal elevation of lipid related indexes in MAD patients who met the inclusion criteria and the upper limit of normal values of alanine aminotransferase (ALT) and aspartate aminotransferase (AST) 2.0 due to long-term stable use of statins were not considered as the basis for exclusion].
6. hepatitis B surface antigen (HBsAg), hepatitis C antibody (HCVAb), syphilis antibody and human immunodeficiency virus (HIV) antibody test are positive at screening.
7. Have gastrointestinal, liver, kidney, or other diseases known to interfere with the absorption, distribution, metabolism, or excretion of drugs.
8. History of drug abuse in the 12 months prior to the first administration of the study drug or alcohol abuse in the 3 months prior.
9. A clinically significant allergic reaction that the investigator believes interferes with the subject's ability to participate in the trial; Known allergies to any of the study drug ingredients.
10. Any live vaccine was administered within 30 days prior to the first administration of the study drug.
11. Pregnant or lactating women.
12. Donate blood or plasma within 3 months prior to the first administration of the study drug, or lose more than 500mL of whole blood, or receive blood transfusion within 1 year prior to the first administration of the study drug.
13. History of Participating in another investigational clinical trial within 90 days before the first administration of the study drug.
14. Any other factors considered by the investigator to be inappropriate for participation in the trial.
15. Additional exclusion criteria for SAD subjects: Use of any prescription and over-the-counter drugs during the 14 days prior to the first administration of the study drug or during the 5 half-lives of the drug, whichever is longer, unless deemed by both the investigator and the sponsor to be of no clinical relevance and not to affect lipid levels.
16. Additional exclusion criteria for MAD subjects:

    1. Use of any prescription and over-the-counter drugs during the 14 days prior to the first administration of the study drug or during the 5 half-lives of the drug, whichever is longer, unless deemed by both the investigator and the sponsor to be of no clinical relevance and not to affect lipid levels.Blood pressure medications (up to 2 blood pressure medications per subject) are permitted, and subjects who are treated with statins are allowed to take a stable dose of simvastatin, atorvastatin or rosuvastatin according to the protocol.
    2. Patients with homozygous familial hypercholesterolemia (HoFH).
    3. Secondary dyslipidemia.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 96 (Actual)
Dates: Start 2022-02-22 (Actual); Primary Completion 2022-09-21 (Actual); Study Completion 2022-12-08 (Actual)

PRIMARY OUTCOMES:
The number and severity of treatment emergent adverse events (TEAEs) . | 5 days after single dose and 18 days after the first dose of multiple doses
  To assess the safety and tolerability of single or multiple oral dose of HSK31679 in healthy or LDL-C elevated adult volunteers
Changes from baseline in clinical laboratory parameters（Blood routine, blood biochemistry, Urine routine, Coagulation function, thyroid function and antibodies）. | 5 days after single dose and 18 days after the first dose of multiple doses
  To assess the safety and tolerability of single or multiple oral dose of HSK31679 in healthy or LDL-C elevated adult volunteers
Changes from baseline in physical examination results（General condition skin mucous membrane superficial lymph nodes head neck chest abdomen spine limbs and others）. | 5 days after single dose and 18 days after the first dose of multiple doses
  To assess the safety and tolerability of single or multiple oral dose of HSK31679 in healthy or LDL-C elevated adult volunteers
Changes from baseline in vital signs（Systolic and diastolic blood pressure, pulse, respiratory rate, body temperature）. | 5 days after single dose and 18 days after the first dose of multiple doses
  To assess the safety and tolerability of single or multiple oral dose of HSK31679 in healthy or LDL-C elevated adult volunteers
Changes from baseline in 12-ECG（QT interval, QTcF interval, PR interval, QRS interval and RR interval）. | 5 days after single dose and 18 days after the first dose of multiple doses
  To assess the safety and tolerability of single or multiple oral dose of HSK31679 in healthy or LDL-C elevated adult volunteers

SECONDARY OUTCOMES:
Plasma concentration of HSK31679 | 0 to 24 hours on Day 1 and Day 14
  Assessed with or without food in single dose Assessed with or without stains in multiple doses
Lipid level changes following administration of HSK31679 | Day 1 to Day 14
  Assessed with or without stains in multiple doses

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Peking University First Hospital, Beijing, Beijing Municipality
  - Xiangya Hospital of Central South University, Changsha